CLINICAL TRIAL: NCT05672342
Title: A Pilot Study to Evaluate the Benefits of Phytocannabinoids for the Treatment of Chronic Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Phytocannabinoids for the Treatment of Chronic Chemotherapy-Induced Peripheral Neuropathy in Breast and Colon Cancer Survivors
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: withdrawn
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22339; NCI-2022-10253 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22339 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH); R21CA260447 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Carcinoma; Chemotherapy-Induced Peripheral Neuropathy; Colon Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms | interventions — Cannabidiol; delta-8-tetrahydrocannabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (CBD) (Experimental): Patients receive CBD PO on study.
  Interventions: Drug: Cannabidiol; Other: Questionnaire Administration
- Arm II (CBD + THC) (Experimental): Patients receive CBD PO + THC PO on study.
  Interventions: Drug: Cannabidiol; Drug: Delta-8-Tetrahydrocannabinol; Other: Questionnaire Administration
- Arm III (placebo) (Placebo Comparator): Patients receive placebo PO on study.
  Interventions: Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cannabidiol — Given PO
  Other Names: CBD; CBD Oil; Epidiolex; GWP42003-P
  Arms: Arm I (CBD); Arm II (CBD + THC)
Drug: Delta-8-Tetrahydrocannabinol — Given PO
  Other Names: .DELTA.8-TETRAHYDROCANNABINOL; delta-8-THC
  Arms: Arm II (CBD + THC)
Drug: Placebo Administration — Given PO
  Arms: Arm III (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well phytocannabinoids (cannabidiol [CBD] and tetrahydrocannbinol [THC]) work in reducing chronic chemotherapy-induced peripheral neuropathy (CIPN) in breast and colon cancer survivors. Neuropathy is the most common neurological symptom reported by cancer patients due to treatment. A variety of pharmacologic treatments have been evaluated to alleviate CIPN symptoms; however, no definitive treatment has been found to successfully treat all the symptoms of CIPN. Therefore, investigators continue to seek other possible treatment options including cannabis. Phytocannabinoids may be a particularly useful intervention for cancer patients given the limited effective treatments for CIPN. In addition, cannabis-based medicines have become tremendously popular as both cancer patients and clinicians are seeking therapies with fewer potential risks of dependency and other side effects. This trial is being done to provide cancer patients and clinicians with reliable information to help guide their use of phytocannabinoids to manage the tremendous distress and pain experienced by many cancer patients, which impacts their long-term quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the ability of CBD and THC:CBD to reduce CIPN symptoms as compared to placebo using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG)-Neurotoxicity (Ntx) subscale among breast and colon cancer survivors.

SECONDARY OBJECTIVES:

I. Evaluate the impact of CBD and THC:CBD as compared to placebo on quality of life using the Functional Assessment of Cancer Therapy General (FACT-G) among breast and colon cancer survivors with chronic CIPN.

II. Document the utilization of neuropathic and pain medications by cancer patients with chronic CIPN during treatment with CBD and THC:CBD as compared to placebo.

III. Describe the side effects of CBD and THC:CBD treatment.

EXPLORATORY OBJECTIVES:

I. Assess neurological symptoms and function with the Neuropathy Pain Scale (NPS), Total Neuropathy Sccore - clinically based (TNSc), quantitative sensory testing (QST), Grooved Pegboard Test (GPT), and Unipedal Stance balance test (USBT) among patients with chronic CIPN treated with CBD and THC:CBD as compared to placebo.

II. Evaluate for predictors of response to CBD and THC:CBD for chronic CIPN.

OUTLINE: This is a dose-escalation study of CBD and THC. Patients are randomized to 1 of 3 arms.

ARM I: Patients receive CBD orally (PO) on study.

ARM II: Patients receive CBD PO + THC PO on study.

ARM III: Patients receive placebo PO on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Willingness to comply with all study interventions including the use of medical cannabis and follow-up assessments
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Ability to read and understand English for questionnaires
* Patients must have either neuropathy >= 1 according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 scale or a neuropathy score of > 3 on a 0-10 scale plus a FACT/GOG-Ntx score of > 10
* The patient's previous chemotherapy treatment must have included a taxane (paclitaxel, nab-paclitaxel, or docetaxel) or platinum (cisplatin, oxaliplatin, or carboplatin) and considered the primary cause of the neuropathy by the medical team
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease)
* Aspartate aminotransferase (AST) =< 3 x ULN
* Alanine aminotransferase (ALT) =< 3 x ULN
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* Current active treatment with chemotherapy, radiation or surgery in the past 3 months or planned treatment during this study protocol period. Note: Hormonal therapy is allowed

Exclusion Criteria:

* Concurrent use of other alternative medicines such as medical cannabis, herbal agents and high dose vitamins and minerals
* Liver cirrhosis Child-Pugh B or C
* Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry (These patients may not be able to cooperate with this slightly invasive procedure or with the data collection process)
* History of diabetic neuropathy, neuropathy related to human immunodeficiency virus (HIV), or other medical causes of chronic neuropathy in the baseline assessment including past medical history, any history of diabetes, alcoholism, and vitamin B deficiency
* Previous medical cannabis use for any indication within 30 days of enrollment
* Planned or actual changes in type of medications that could affect symptoms related to CIPN. New medications for the treatment of CIPN are not allowed during the study.

  * Note: Subjects need to be on stable doses of CIPN medications for 4 weeks
* Strong inhibitors or inducers of CYP3A4
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Diagnosis of Gilbert's disease
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-06 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG)-Neurotoxicity (Ntx) subscale scores | Baseline up to week 12
  The primary analysis will compare difference in scores from the FACT/GOG-Ntx between all groups using analysis of variance, and a repeated measures analysis of variance analysis will be performed. Multivariable mixed-effects regression model which takes possible dependence of longitudinal measurements within each subject into account, will be used. In addition, a paired t-test will be utilized to compare scores between baseline and 8 and 12 weeks of treatment for each group separately.

SECONDARY OUTCOMES:
Quality of life by the Functional Assessment of Cancer Therapy-General (FACT-G) scores | Up to 12 weeks
  The pre-treatment values recorded from the FACT-G will be considered the baseline scores. A paired T-test will be utilized to compare scores between baseline and 8 weeks of treatment. For comparisons between groups at four specific assessment points (baseline, week 4, week 8, and week 12), a repeated measures analysis of variance analysis will be performed
Utilization of neuropathic and pain medications | Up to 12 weeks
  Medication data will initially be analyzed as a dichotomous variable (yes/no) for each medication. These medications may include neuropathic medications (e.g., gabapentin, pregabalin, duloxetine, amitriptyline), Non-steroidal anti-inflammatory drugs, acetaminophen, opioid medications (e.g., morphine, oxycodone), or other related medications. Comparisons between the baseline and after-treatment medication status will be analyzed using McNemar's test. Including all the time points in the analysis of any single medication will use Cochran's Q test. The usage of multiple medications will be summarized descriptively to determine the best way to quantify multiple use, such as counts or categorized quantities. McNemar's test will be used to detect change in the level of medication use.
Incidents of adverse events | Up to 12 weeks
  All adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 6.0. The severe adverse events (SAE) (grade >= 3) will be tabulated per treatment arm and the difference of SAE will be compared among groups using chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lee, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States